CLINICAL TRIAL: NCT00710164
Title: Effectiveness and Safety of Xiaoshuanchangrong (XSCR) Capsule for the Treatment of Patients Who Have Suffered From a Stroke
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Collaborators: Sizuo (Unknown)
Responsible Party: Dr. Cai, Department of Integrative Medicine, Zhongshan hospital, Fudan University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XSCR capsule-1
Record Dates: First submitted 2008-07-01; First posted 2008-07-04 (Estimated); Last update posted 2010-05-28 (Estimated); Status verified 2009-09

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Honghua extract, Carthamus tinctorius

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental)
  Interventions: Drug: XSCR capsule (Composed of Traditional Chinese Medicine Huangqi, Chuanxiong, Chishao, Danggui, Dilong, Taoren, Honghua.)
- B (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: XSCR capsule (Composed of Traditional Chinese Medicine Huangqi, Chuanxiong, Chishao, Danggui, Dilong, Taoren, Honghua.) — 14 days of XSCR capsule
  Arms: A
Drug: Placebo — 14 days of Placebo
  Arms: B

SUMMARY:
This study will determine if Xiaoshuanchangrong (XSCR) capsule will improve recovery from an acute stroke. The study is designed to look at both overall recovery and recovery of motor function, for example muscle strength and coordination.

ELIGIBILITY:
Inclusion Criteria:

* Acute ischemic stroke with limb weakness, NIH stroke scale ≥6, limb weakness score ≥2
* Onset of symptoms within 72 hours
* 18 Years and older
* Consistent with the Qi deficiency and Blood stasis type by Traditional Chinese Medicine (TCM) standard
* Patients or their representatives voluntarily take part in this study and signed the informed consent

Exclusion Criteria:

* Transient ischemic attack(TIA), cerebral hemorrhage, subarachnoid hemorrhage
* Subjects who are unlikely to complete taking the investigational product and/or are unlikely to undergo active medical management during that period due to a severe clinical condition.
* Pregnant or breast-feeding.
* Proven disability by law, such as blindness, deafness, dumb, disturbance of intelligence, mental disorders, limb handicap.
* Liable to be allergic (allergic to at lease 2 foods/drugs previously exposed)
* Had been participated in other clinical trials during the last 1 month prior to study inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2008-09; Primary Completion 2010-07 (Estimated)

PRIMARY OUTCOMES:
Global disability on modified Rankin scale | 90 days

SECONDARY OUTCOMES:
NIH stroke scale | 90 days
Barthel Index | 90 days
Syndrome score by Traditional Chinese Medicine (TCM) standard | 90 days
mini-mental state examination (MMSE) | 90 days
Changes in laboratory indexes as safety assessment, including red blood cell(RBC), white blood cell(WBC), platelet(PLT), alanine transaminase (ALT), aspartate transaminase(AST), blood urea nitrogen (BUN), creatinine(Cr) in blood samples; protein, red b | 90 days

CONTACTS AND LOCATIONS:
Locations (20):
- China (20):
  - Department of Nuerology, Kunming General Hospital of Chengdu Military Command, Kunming, Chengdu
  - Department of Nuerology, The Second People's Hospital of Foshan city, Foshan, Guangdong
  - Department of Nuerology, The Second People's Hospital of Jiangmen city, Jiangmen, Guangdong
  - Department of Nuerology, Liuzhou Hospital of Traditional Chinese Medicine, Liuchow, Guangxi
  - Department of Nuerology, Cangzhou Central Hospistal, Cangzhou, Hebei
  - Department of Nuerology, Hubei Hospital of Traditional Chinese Medicine, Wuhan, Hubei
  - Department of Nuerology, The First People's Hospital of Changsha city, Changsha, Hunan
  - Department of Neurology, Renji Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Department of Nuerology, Changzheng Hospital Affiliated to the Second Military Medical University, Shanghai, Shanghai Municipality
  - Department of Integrative Medicine, Zhongshan hospital, Fudan University, Shanghai, Shanghai Municipality
  - Department of Nuerology, Shuguang Hospital Affiliated to Shanghai University of Traditional Chinese Medicine, Shanghai, Shanghai Municipality
  - Department of Neurology, Ruijin Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Department of Nuerology, Longhua Hospital Affiliated to Shanghai University of Traditional Chinese Medicine, Shanghai, Shanghai Municipality
  - Department of Nuerology, Zhongshan hospital, Fudan University, Shanghai, Shanghai Municipality
  - Department of Neurology, Huashan hospital, Fudan University, Shanghai, Shanghai Municipality
  - Department of Nuerology, Tongji Hospital of Tongji University, Shanghai, Shanghai Municipality
  - Department of Neurology, Shanghai First People's Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Department of Nuerology, Xinhua Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Department of Nuerology, Shanghai Sixth People's Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Department of Neurology, Changhai Hospital Affiliated to the Second Military Medical University, Shanghai, Shanghai Municipality